CLINICAL TRIAL: NCT05610592
Title: Prognostic Impact of Tumor Budding and Tumor-infiltrating Lymphocytes in Patients With Colorectal Cancer Under Different MMR Status: A Single-Center, Open-Label, Retrospective, Observational Cohort Study
Brief Title: Tumor Budding in Patients With Colorectal Cancer Under Different MMR Status
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Other Study IDs: GIHSYSU-31
Record Dates: First submitted 2022-11-04; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Tumor Budding; Rectal Cancer
Keywords: Tumor budding; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rectal cancer: patients underwent curative surgery
  Interventions: Procedure: total mesorectal exicision

INTERVENTIONS:
Procedure: total mesorectal exicision

SUMMARY:
This study investigates the ability of tumor budding to identify prognosis in different MMR states and different levels of tumor lymphocyte infiltration. Tumor budding is usually defined as an isolated single cancer cell or a cluster of up to four cancer cells located at the front of an infiltrating tumor.

DETAILED DESCRIPTION:
As a component of the tumor microenvironment, tumor budding is associated with the epidermal mesenchymal transition of tumor cells and may predict disease progression and poor survival. The current assessment of tumor budding levels is mainly based on the ITBCC grading system. The dMMR phenotype of colorectal cancer is associated with the generation of non-self-recognizing neoantigens by the immune system, with tumor-associated extensive inflammatory cell infiltration, and often the dMMR phenotype of colorectal cancer has a lower level of outgrowth, possibly with the generation of local immune responses capable of eradicating tumor budding cells. The prognostic value of the conventional tumor budding grading system has been validated mainly in stage I and II colorectal cancers and does not consider the effect of MMR status on tumor budding. This retrospective study is designed to investigate whether the high grade of tumor budding under high immune response status implies immune escape of tumor cells and brings worse survival outcome, establish a more independent risk grading system to maximize the prognostic value of tumor budding in dMMR phenotype of colorectal cancer in combination with tumor-infiltrating lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed colorectal adenocarcinoma cancer pathologically
2. Underwent primary surgery
3. With records for tumor budding staining
4. Willing and able to provide written informed consent for participation in this study
5. Non-complicated primary tumor (complete obstruction, perforation, bleeding)

Exclusion Criteria:

1. With distant metastases at the time of initial diagnosis
2. Without a complete pathological date
3. Hereditary colorectal cancer
4. Subjects with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients underwent curative surgery
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
5-year event-free survival rate | 5 years after the surgery

SECONDARY OUTCOMES:
5-year overall survival rate | 5 years after the surgery
Local recurrence | 5 years after the surgery
  Defined as an intrapelvic recurrence following a primary rectal cancer resection, with or without distal metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous information may be provided upon reasonable request